CLINICAL TRIAL: NCT01636115
Title: Validation of Muscle Strength Testing for Pectoralis Major
Status: Completed | Type: Observational
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Hsin-Min Lee, Associate Professor, National Science and Technology Council, Taiwan
Other Study IDs: ISU-IRB-101-001
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Pectoralis Major; Muscle Strength; Surface EMG; Force Measurement

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

SUMMARY:
This study wants to understand which direction of shoulder movement and what posture of shoulder are best for the procedure of muscle strength testing of the muscle pectoralis major(PM). We will use muscle activity signals (sEMG) and force measurement to analyze the contribution of two parts of PM in three different contraction direction with three different shoulder postures.

ELIGIBILITY:
Inclusion Criteria:

* Young male subjects which could expose the area of anterior chest to paste the sEMG electrodes

Exclusion Criteria:

* Injury and uncomforted one week before the test

Ages: 17 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Students in University.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
sEMG | 6/1/2012
  Surface EMG signal were collected.

CONTACTS AND LOCATIONS:
Locations (1):
- I-Shou university, Kaohsiung City, Taiwan